CLINICAL TRIAL: NCT00562003
Title: A Phase I Study of a Tropism Modified Conditionally Replicative Adenovirus Vector (Ad5-Delta 24 RGD)for Intraperitoneal Delivery in Ovarian and Extraovarian Cancer Patients (Infectivity Enhanced Virotherapy for Ovarian Cancer)
Brief Title: Safety Study of a Genetically Modified Adenovirus in Ovarian Cancer Patients
Acronym: Ad5Delta24RGD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ronald D. Alvarez, MD / Director,Division of Gynecologic Oncology, UAB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F061005016 (UAB 0643); UAB 0643
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer
Keywords: Ovarian cancer study
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Tenckhoff Catheter placement — 'Tenckhoff catheter' will be placed into the abdominal cavity by a minor surgical procedure performed in the Radiology Department.
Drug: Ad5-delta24RGD — Within two weeks before the start of the study, a physical exam, blood tests, removal of fluid from abdominal cavity through the catheter and a CT scan of abdomen and pelvis will be performed.
  The procedure will involve receiving the Ad5-delta24RGD virus once a day for 3 days. The virus will be put into the abdominal cavity through a 'Tenckhoff catheter'.

SUMMARY:
The primary purpose of this study is to determine the maximally tolerated dose and spectrum of toxicities encountered with intraperitoneal delivery of a RGD modified conditionally replicative adenovirus (Ad5-Delta 24RGD) in patients with recurrent ovarian cancer.

Secondary objectives :

* To determine the biologic effects encountered with intraperitoneal delivery of Ad5-Delta 24RGD in patients with recurrent ovarian cancer cells
* To determine immunologic response generated against Ad5-Delta 24RGD when administered intraperitoneally to patients with recurrent ovarian adenocarcinoma
* To determine potential clinical activity of Ad5-Delta 24RGD when administered intraperitoneally to patients with recurrent ovarian adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented invasive epithelial ovarian or extra-ovarian adenocarcinoma
* Patients must have persistent or recurrent disease after standard debulking/staging surgery and conventional chemotherapy.Prior chemotherapy must have included a taxane/platinum based regimen
* Patients must have evidence of intraabdominal disease; disease may be measurable or nonmeasurable
* Patients must have a GOG performance status of 0, 1, or 2, and have a life expectancy of greater than 3 months
* Patients must have adequate hematologic, renal, cardiac, pulmonary, coagulation, and hepatic function defined as:

  1. WBC> 3,000 ul
  2. Granulocytes> 1,500 ul
  3. Platelets> 100,000
  4. Creatinine clearance (actual or calculated) >80 mg/dl or serum creatinine <2.0
  5. Serum transaminases <2.5x upper limits of normal
  6. Normal serum bilirubin
  7. PT/PTT/INR < 1.5 x institutional ULN
  8. Ejection fraction on echocardiogram > 55%
  9. O2 saturation > 92%
* Patients must be 19 years or older (as mandated by Alabama state law) and must have signed informed consent

Exclusion Criteria:

* Patients with epithelial ovarian tumors of low malignant potential (with or without invasive implants), with ovarian stromal tumors, or with germ cell tumors of the ovary are ineligible to participate in the study
* Patients with the only site of disease located beyond the abdominal cavity are ineligible to participate in the study
* Patients who are pregnant or lactating are ineligible to participate in the study
* Patients with a GOG performance status of 3 or 4 are ineligible to participate in the study
* Patients with active heart disease (characterized by angina, unstable arrhythmia, congestive heart failure or EF < 55%, pulmonary hypertension), active or chronic debilitating pulmonary disease (i.e., active pneumonia, severe COPD, pulmonary edema, O2 saturation < 92%), or coagulation disorders (i.e., bleeding disorders, on therapeutic anti-coagulants)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerated dose and spectrum of toxicities of Ad5-Delta24RGD | 1 month

SECONDARY OUTCOMES:
To determine biologic, immunologic, and anti-tumor effects of Ad5-delta24RGD | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Alvarez, M.D., Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- UAB Highlands, 1201 11th Ave S, 4th Floor, Gynecologic Oncology, Birmingham, Alabama, United States